CLINICAL TRIAL: NCT03765281
Title: Exploring the Outcomes of System Supports for Youth With Mental Illness and/or Addictions and Their Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Anthony Levitt, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 040-2018
Record Dates: First submitted 2018-06-28; First posted 2018-12-05 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Mental Health Disorder; Addiction
MeSH Terms: conditions — Mental Disorders; Behavior, Addictive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Navigation (Experimental): Navigation intervention plus Resource List
  Interventions: Other: Navigation; Other: Resource List
- Self-Navigation (Active Comparator): Resource List intervention
  Interventions: Other: Resource List

INTERVENTIONS:
Other: Navigation — Service delivered by clinical Navigator who learns about youth and family's needs and matches to appropriate services.
  Arms: Navigation
Other: Resource List — Extensive list of mental health and addictions resources, information, and services. Contact information and web links provided for individuals to explore and contact resources of interest.

SUMMARY:
This trial (Phase II) will assess the different methods of supporting families in finding mental health and/or addictions (MHA) services for youth. Youth with MHA issues and their families are particularly vulnerable in the MHA system, due to a lack of specialized support and complicated transitions between services. This study will assess the potential impact of Navigation on youth MHA symptom reduction or functional improvement, family functioning, satisfaction with MHA services, as well as the cost-benefit of Navigation. This project will seek to determine whether there is a difference for those youth with MHA issues and their families who receive Navigation over those who find and access MHA care on their own.

DETAILED DESCRIPTION:
This pilot feasibility trial (Phase I) assessed the feasibility to conduct a randomized controlled trial examining whether families of youth ages 13 to 26 with mental illness and/or addiction concerns who receive Navigation services experience improved clinical outcomes compared to families who interact with the MHA care system on their own (usual care). This pilot feasibility trial (Phase I) assessed the different methods of supporting families in finding mental health and/or addictions (MHA) services for youth. Youth with MHA issues and their families are particularly vulnerable in the MHA system, due to a lack of specialized support and complicated transitions between services. This study assessed the potential impact of Navigation on youth MHA symptom reduction or functional improvement, family functioning, satisfaction with MHA services, as well as the cost-benefit of Navigation and sought to determine whether there is a difference for those youth with MHA issues and their families who receive Navigation over those who find and access MHA care on their own.

The primary outcomes for Phase I of this trial were:

1. Recruitment rate as a measure of recruitment feasibility (baseline): tracking of recruitment rate to determine whether it is high enough for a full-scale trial to be feasible.
2. Change in acceptability of study methods across time (two months and four months): Acceptability of Procedures and assessments by participants as measure of protocol feasibility (Questionnaire developed based on the Theoretical Framework of Acceptability, Sekhon et al., 2017).
3. Study Completion Rate (four months): tracking of study completion rate to determine whether it is high enough for a full-scale trial to be feasible.

The secondary outcomes for Phase I of this trial were:

1. Caregiver Strain Across Time (baseline, two months, four months): Caregiver Strain Questionnaire as measure of functional and health outcomes for the youth and family (CSQ; Bickman et al., 2012). Clinical Outcome #1.
2. Youth Symptoms & Functioning Across Time (baseline, two months and four months): Symptoms and Functioning Severity Scale (SFSS, Bickman et al., 2012).Clinical Outcome #2.Total Scale Range= Min: 26, Max: 130. Higher values = worst outcome.
3. Family Functioning Across Time (baseline, two months and four months) (baseline, two months and four months): Olson Family Satisfaction Scale (FSS, Olson, 2010). Clinical Outcome #3. Total Scale range = Min: 10, Max: 50. High values = better outcome.
4. Youth Emotion & Behaviour Symptoms Across Time (baseline and four months): Child and Adolescent Symptom Inventory (CASI, Sprafkin et al., 2010). Clinical Outcome #4. Total Scale Range = Min 29, Max: 87. Higher values = worst outcome.
5. Caregiver Quality of Life Across Time (baseline and four months): Medical Outcomes Survey Short-Form (SF-36, RAND Health, 2018). Clinical Outcome #5. Total Scale Range = Min: 36, Max: 180. Higher values = worst outcome.
6. Youth Quality of Life Across Time (baseline and four months): Medical Outcomes Survey Short-Form (SF-36; RAND Health, 2018). Clinical Outcome #6. Total Scale Range = Min: 36, Max: 180. Higher values = worst outcome.

Other outcome measures:

1. Health Services Utilization over time (baseline and four months): Health Services Utilization Questionnaire (Henderson et al., 2017) Reporting of usage of health services for purposes of cost change estimates.
2. Health Services Utilization over time (baseline and four months): Child and Adolescent Services Assessment (CASA; Ascher et al., 1996); Reporting of access of health services for services usage estimates.

ELIGIBILITY:
Inclusion Criteria:

* family member of youth age 13 to 26 who is experiencing a mental health concern and/or substance use issue
* residing in the Greater Toronto Area
* seeking mental health and/or addictions services or supports

Exclusion Criteria:

* currently in crisis
* previously received navigation support at Sunnybrook Health Sciences Centre.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
Caregiver Strain Across Time | Change in Caregiver Strain from baseline to twelve months
  Caregiver Strain Questionnaire as measure of functional and health outcomes for the youth and family (CSQ; Bickman et al., 2012); Clinical Outcome #1. Total Scale Range= Min: 7, Max: 35. Higher scores: worst outcome.
Youth Symptoms & Functioning Across Time | Change in Youth Functioning from baseline to twelve months
  Symptoms and Functioning Severity Scale (SFSS, Bickman et al., 2012); Clinical Outcome #2. Total Scale Range= Min: 26, Max: 130. Higher scores = worst outcome.
Family Functioning Across Time | Change in Family Functioning from baseline to twelve months
  Olson Family Satisfaction Scale (FSS, Olson, 2010); Clinical Outcome #3. Total scale range = Min: 10, Max: 50. Higher scores = better outcome.
Caregiver Quality of Life Across Time | Change in Caregiver Quality of Life from baseline to twelve months
  World Health Organization Quality of Life Instruments (WHOQOL-BREF Field Trial Version, WHOQOL Group, 1991); Clinical Outcome #4. Total Scale Range = Min: 4, Max: 20. High scores = better outcome.
Youth Quality of Life Across Time | Change in Youth Quality of Life from baseline to twelve months
  Kid - & Kiddo-KINDL Parent's Questionnaire KINDL Quality of Life Questionnaire for Children (Kid- & Kiddo-KINDL, Ravens-Sieberer & Bullinger, 2000); Clinical Outcome #5. Total Scale Range = Min: 24, Max: 120. High scores = better outcome.

OTHER OUTCOMES:
Health Services Utilization Questionnaire over time | Change in Health Services Utilization from baseline to twelve months
  Health Services Utilization Questionnaire (Henderson et al., 2017) Reporting of usage of health services for purposes of cost change estimates.
Health Services Satisfaction Questionnaire | Change in Health Services Satisfaction from baseline to twelve months
  Reporting of satisfaction with health services accessed.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Levitt, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No